CLINICAL TRIAL: NCT07348393
Title: A Phase 2, Single Arm Multicenter, Study Testing Mezigdomide, Carfilzomib, and Dexamethasone (480Kd) in Participants With Relapsed or Refractory Multiple Myeloma (RRMM)
Acronym: Mezi-KD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP241725
Record Dates: First submitted 2025-12-19; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Relapsed or Refractory Multiple Myeloma (RRMM)
Keywords: Relapsed or Refractory Multiple Myeloma (RRMM); Mezigdomide; Carfilzomib; Dexamethasone
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (single arm) (Experimental): Administration of a combination of treatments : Mezigdomide / Carfilzomib / Dexamethasone
  Interventions: Drug: Administration of a combination of treatments

INTERVENTIONS:
Drug: Administration of a combination of treatments — Administration of a combination of treatments : Mezigdomide / Carfilzomib / Dexamethasone

SUMMARY:
Despite advances in multiple myeloma (MM) therapy, patients continue to suffer from frequent relapses and treatment-resistant disease. Therefore, additional novel, safe, and effective therapies are needed to drive deeper and more prolonged responses for patients with RRMM.

Mezigdomide (also known as CC-92480 or BMS-986348) is a novel, highly potent cereblon (CRBN)-E3 ligase modulating drug (CELMoD) and represents a new generation of CRBN-modulating (CM) agents optimized to induce rapid and robust degradation of the transcription factors Aiolos and Ikaros, which are important regulators for lymphocyte development and differentiation. CC-92480 was discovered via characterization of structure-activity relationships and exhibits enhanced autonomous cell killing activity in MM cells compared to lenalidomide and pomalidomide due to its increased efficiency at inducing Aiolos and Ikaros degradation. The increased potency of Mezigdomide (also overcomes lenalidomide and pomalidomide resistance in preclinical models inducing potent antiproliferative activity and apoptosis in MM cells with acquired resistance to lenalidomide or pomalidomide.

Carfilzomib is a selective PI that irreversibly binds the proteasome, eliciting antimyeloma activity through unfolded protein stress response and other mechanisms. Carfilzomib is indicated for the treatment of RRMM in combination with dexamethasone (Kd), lenalidomide plus dexamethasone (KRd), and with anti-CD38 monoclonal antibodies daratumumab and isatuximab plus dexamethasone (DKd and IsaKd). However, as lenalidomide has become the foundation for a wide range of regimens used in newly diagnosed multiple myeloma (NDMM) and early in the therapeutic course of MM, KRd is not always a relevant therapeutic option in RRMM. In addition, given the increasing use of anti-CD38 mAb therapy in NDMM and early lines of therapy, DKd and IsaKd will also become less attractive therapeutic options in RRMM. This study will explore mezigdomide with carfilzomib and dexamethasone (480Kd) in a patient population where KRd and DKd/IsaKd are not appropriate treatment options due to prior treatment with lenalidomide and anti-CD38 mAb therapy.

Mezigdomide has shown marked synergy in combination with PIs in lenalidomide resistant mouse xenograft models with combination treatment resulting in near complete tumor regressions. The combination of mezigdomide with carfilzomib has also shown synergistic anti-proliferative activity in MM cell lines resistant to lenalidomide and deeper tumor cell killing than combinations of other

CELMoD agents with carfilzomib. These preclinical data demonstrate the potent synergy of mezigdomide with PIs, including carfilzomib, and the ability of mezigdomide to overcome IMiD drug resistance.

The pleiotropic anti-myeloma effects of mezigdomide include its potent tumoricidal activity in IMiD (lenalidomide and pomalidomide)-resistant cell lines, synergistic anti-tumor effects when combined with proteasome inhibitors and dexamethasone, and the promising clinical activity seen in the Phase 1/2 CC-92480-MM-002 study, all make 480Kd a highly attractive regimen to be further investigated for the treatment of RRMM patients.

This study is a single arm multicenter, Phase 2 study investigating the efficacy and safety of 480Kd in participants with RRMM who received at least 1 prior line of therapy, including lenalidomide and an anti-CD38 mAb, however are carfilzomib naïve.

DETAILED DESCRIPTION:
This is a Phase 2, single arm national multicenter study. Patients with relapsed/refractory symptomatic multiple myeloma (MM) who meet all inclusion criteria, will receive:

* mezigdomide 1 mg on days 1-21 of 28-day cycle, plus
* carfilzomib 20 mg/m2 on day 1 and 56 mg/m2 on day 8, 15 in cycle 1, subsequently 56 mg/m2 on day 1, 8, 15 in cycles 2-12, subsequently 56 mg/m2 on day 1, 15 from cycles 13, plus
* dexamethasone: 40mg (20mg for ≥75yr) on day 1, 8, 15, 22 Patients will be followed according to standard of care and disease will be evaluated on day 1 of each of 28-day cycles of treatment (usually 28 days cycle). Treatment will be continued according to standard practice until MM relapse/progression or toxicity. In case of treatment discontinuation, disease response will still be monitored monthly.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent
2. Adult patients (≥18 years old)
3. ECOG Performance Status score of 0, 1, or 2.
4. Participant has documented diagnosis of multiple myeloma (MM) and measurable disease, defined as any of the following:

   1. M-protein ≥ 0.5 g/dL by serum protein electrophoresis (sPEP), or
   2. M-protein ≥ 200 mg/24-hour urine collection by urine protein electrophoresis (uPEP) or,
   3. For participants without measurable disease in sPEP or uPEP: serum free light chain (sFLC) levels > 100 mg/L (10 mg/dL) involved light chain and an abnormal κ/λ FLC ratio.
5. Participant has received one or two prior line of anti-myeloma therapy. Note: One line can contain several phases (eg, induction, [with or without] hematopoietic stem cell transplant, (with or without) consolidation, and/or [with or without] maintenance therapy).
6. Participant must have received prior treatment with lenalidomide and an anti-CD38 monoclonal antibody.
7. Participant achieved minimal response [MR] or better to at least 1 prior anti-myeloma therapy.
8. Participant must have documented disease progression during or after their last antimyeloma regimen.
9. Reproductive Status

   • Females of childbearing potential (FCBP) must :
   * Have 2 negative pregnancy tests as verified by the Investigator prior to starting study therapy and must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the participant practices true abstinence* from heterosexual contact.
   * Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, 2 forms of contraception: one highly effective, and one additional effective (barrier) contraception without interruption, 28 days prior to starting study intervention, during treatment (including dose interruptions), and for at least 28 days after the last dose of CC-92480, or 6 months after the last dose carfilzomib, whichever is longest.

   Refer to the Celgene CC-92480/BMS-986348 Pregnancy Prevention Plan for additional guidance.

   Note: A FCBP is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy or amenorrhea due to other medical reasons does not rule out childbearing potential) for at least 24 consecutive months (eg, has had menses at any time in the preceding 24 consecutive months).

   • Male participants must :

   - Practice true abstinence* (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a FCBP while participating in the study, during dose interruptions and for at least 90 days after the last dose of CC-92480 or carfilzomib, even if he has undergone a successful vasectomy.

   Refer to the Celgene mezigdomide Pregnancy Prevention Plan for additional guidance.

   * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (eg, calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   * Male participants must agree to refrain from donating sperm while on study intervention, during dose interruptions, and for at least 90 days following last dose of mezigdomide or carfilzomib.
   * Females must agree to refrain from donating eggs while on study intervention and for at least 28 days after last dose of mezigdomide
   * Participants must agree to refrain from donating blood while on study intervention, during dose interruptions, and for at least 28 days following the last dose of study intervention.
   * All male and female participants must follow all requirements defined in the Pregnancy Prevention Plan in Appendix 11 for mezigdomide

   Exclusion Criteria:
   * Participant that received > 3 prior line of anti-myeloma therapy.
   * Medical conditions

     * Participant who has had prior treatment with mezigdomide or carfilzomib.
     * Participant who has had any investigational agents within 28 days or 5 half-lives (whichever is shorter) of initiating study intervention (Participation in another interventional clinical trial concurrent with this study is not permitted, except for those who have completed treatment with the prior investigational agent(s) and are currently in long-term follow-up.)
     * Participant has received any of the following:
   * Plasmapheresis within the last 28 days of initiating study intervention.
   * Major surgery (as defined by the Investigator) within 28 days of initiating study intervention.
   * Radiation therapy, other than local palliative therapy, for myeloma-associated bone lesions within 14 days of initiating study intervention.
   * Use of any systemic anti-myeloma drug therapy within 14 days of initiating study intervention.

     * Participant has previously received allogeneic stem cell transplant at any time or received autologous stem cell transplant within 12 weeks of initiating study treatment.
     * Participant has plasma cell leukemia, Waldenstrom macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or clinically significant light-chain amyloidosis.
     * Participant with known central nervous system (CNS) involvement with myeloma.
     * Participant has any significant medical condition, including active or uncontrolled infection, presence of laboratory abnormality, or psychiatric illness that places the participant at an unacceptable risk for treatment-related complications, if he/she were to participate in the study.
     * Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 14 days for mild or asymptomatic infections or 28 days for severe/critical illness prior to initiating study intervention (Acute symptoms must have resolved and there are no sequelae that would place the participant at a higher risk of receiving study intervention, based on Investigator assessment in consultation with the Sponsor Medical Monitor)
     * Participant has any condition that confounds the ability to interpret data from the study
     * Participant has any of the following laboratory abnormalities:
   * Absolute neutrophil count (ANC) < 1,000/¬µL. It is not permissible to administer GCSF to achieve minimum ANC levels within 7 days prior to screening complete blood count (CBC) (or within 14 days prior for pegfilgrastim).
   * Platelet count: < 75,000/¬µL for participants in whom < 50% of bone marrow nucleated cells are plasma cells; or a platelet count < 50,000/¬µL for participants in whom 'â• 50% of bone marrow nucleated cells are plasma cells. Platelet transfusions are not permitted within 7 days prior to screening complete blood count (CBC).
   * Hemoglobin < 8 g/dL (< 4.9 mmol/L).
   * Estimated glomerular filtration rate (eGFR) < 30 mL/min or requiring dialysis. eGFR will be calculated using the Modification of Diet in Renal Disease (MDRD) formula (see http://mdrd.com).
   * Corrected serum calcium > 13.5 mg/dL (> 3.4 mmol/L)
   * Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5xx upper limit of normal (ULN)
   * Serum total bilirubin > 1.5 x ULN; > 3.0 mg/dL is allowed for participants with documented Gilbert's syndrome.

     * Participant with gastrointestinal disease or surgery (eg, gastric bypass surgery) that may significantly alter the absorption of Mezigdomide and/or other oral study intervention.
     * Participant has prior history of malignancies, other than MM, unless the participant has been free of the disease for 'â• 5 years with the exception of the following noninvasive malignancies:
   * Basal cell carcinoma of the skin
   * Squamous cell carcinoma of the skin in situ (Stage 0)
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is curative

     * Participant has received immunosuppressive medication within the last 14 days of initiating study intervention. The following are exceptions to this criterion:
   * Intranasal, inhaled, or topical corticosteroids or local corticosteroid injections (eg, intra-articular injection).
   * Systemic corticosteroids at doses that do not exceed 10 mg/day of prednisone or the equivalent (see Table 7.7.2-1).
   * Steroids as premedication for hypersensitivity reactions (eg, computed tomography [CT] scan premedication).

     - Administration of strong CYP3A modulators; administration of proton-pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, pantoprazole, rabeprazole) within 2 weeks of starting study intervention.

     - Participant has impaired cardiac function or clinically significant cardiac disease, including any of the following:
   * Myocardial infarction within 1 year before inclusion, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure New York Heart Association Class III-IV) or pericardial disease.
   * Uncontrolled cardiac arrhythmia or clinically significant electrocardiogram (ECG) abnormalities, including prolongation of QT interval on Screening ECG as defined by a QTc interval > 470 msec using Fridericia's QT correction formula
   * Left ventricular ejection fraction < 40% as assessed by transthoracic echocardiogram (TTE) or multigated acquisition scan (MUGA)

     - Participant has uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment.

     - Participant who has had a live vaccine within 3 months of start of study therapy.
     * Participant is unable or unwilling to undergo protocol required thromboembolism or antiviral prophylaxis
     * Participant is positive for human immunodeficiency virus (HIV), chronic or active hepatitis B, active hepatitis A, or active hepatitis C:
   * Known positive HIV status.
   * Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Participants with resolved infection (ie, participants who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. EXCEPTION: Participants with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination do not need to be tested for HBV DNA by PCR.
   * Known to be seropositive for hepatitis C virus (HCV); anti-HCV antibody positive or HCV- ribonucleic acid (RNA) quantitation positive, except in the setting of a sustained virologic response (SVR), defined as viremia at least 12 weeks after completion of antiviral therapy.
   * Reproductive Status

     - Participant is a female who is pregnant or breastfeeding, or who intends to become pregnant during participation in the study.
   * Contraindication to investigational medicinal products (mezigdomide, carfilzomib and dexamethasone)
   * Participation in another interventional study or being in the exclusion period at the end of a previous study.
   * Prior/Concomitant Therapy

     - Inability to comply with restrictions and prohibited treatments as listed in Section 7.7: Concomitant Therapy.
   * Physical and Laboratory Test Findings - Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with the target population
   * Allergies and Adverse Drug Reaction

     * Participant has a history of anaphylaxis or hypersensitivity to thalidomide, lenalidomide (including 'â• Grade 3 rash during prior thalidomide or lenalidomide therapy), carfilzomib or dexamethasone or the excipients contained in the formulations, or participant has any contraindications per local prescribing information.
   * Other Exclusion Criteria - Prisoners or participants who are involuntarily incarcerated. (Note: Under certain specific circumstances and only in countries where local regulations permit, a person who has been imprisoned may be included or permitted to continue as a participant. Strict conditions apply, and BMS approval is required.) - Participants must agree to refrain from donating blood while on study intervention, during dose interruptions, and for at least 28 days following the last dose of study intervention.

   Eligibility criteria for this study have been carefully considered to ensure the safety of the study participants and that the results of the study can be used. It is imperative that participants fully meet all eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Determine the progression-free survival (PFS) of mezigdomide, carfilzomib and dexamethasone (480Kd) in participants with relapsed or refractory multiple myeloma (RRMM) | 2 years
  PFS defined as the time from inclusion to first documentation of progressive disease (PD) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | At 2-years
  Defined as the time from inclusion to time of death due to any cause
Best overall Response Rate (ORR) | 2 years
  Defined as the percentage of participants who achieve best response of partial response (PR) or better according to the IMWG Uniform Response Criteria for Multiple Myeloma
Rate of very good partial response (VGPR) or better (VGPRR) | 2 years
  Defined as the percentage of participants who achieve best response of VGPR or better according to the IMWG Uniform Response Criteria for Multiple Myeloma
Rate of complete response (CR) or better (CRR) | 2 years
  Defined as the percentage of participants who achieve best response of CR or better according to the IMWG Uniform Response Criteria for Multiple Myeloma
Time to Response (TTR) | 2 years
  Defined as the time from inclusion on to the first documentation of response (PR or better)
Duration of Response (DOR) | 2 years
  Defined as the time from the first documentation of response (PR or better) to the first documentation of progressive disease (PD) or death due to any cause, whichever occurs first
Time to Progression (TTP) | 2 years
  Defined as the time from inclusion to the first documentation of PD
Time to Next Treatment (TTNT) | 2 years
  Defined as the time from inclusion to the start of the next anti-myeloma treatment
To evaluate minimal residual disease (MRD) negativity rate in participants treated with 480Kd | 2 years
  the proportion of participants who achieve CR or better and are MRD negative (defined at a sensitivity of a minimum of 1 in 105 nucleated cells)
To evaluate safety of 480Kd in participants with RRMM | 2 years
  Defined as the type, frequency, seriousness and severity of adverse events (AEs), and relationship of AEs to study treatment
To evaluate cancer and multiple myeloma-related symptoms | 2 years
  Using the European Organization for Research and Treatment of Cancer - Quality of Life C30 questionnaire (EORTC QLQ-C30) and the European Quality of Life Multiple Myeloma module (EORTC QLQ-MY20) in participants treated with 480Kd
To evaluate health-related quality of life (HRQoL) | 2 years
  Using HRQoL questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Antoine Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided